CLINICAL TRIAL: NCT00589953
Title: High-Dose Erythropoietin in Very Low Birth Weight Infants for the Potential Treatment of Prematurity-Related Cerebral Hemorrhagic-Ischemic Injury: A Phase II Safety/Tolerability Study
Brief Title: High-Dose Erythropoietin in Extremely Premature Infants to Prevent/Attenuate Brain Injury: A Phase II Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R06-04-004; IND12537
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Infant, Premature; Erythropoietin; Brain Injury; Intraventricular Hemorrhage; Periventricular Leukomalacia; Neurodevelopmental Outcomes; Randomized Clinical Trial
Keywords: Extreme Prematurity; Erythropoietin; Perinatal Brain Injury; Intraventricular Hemorrhage; Periventricular Leukomalacia; Neurodevelopmental Outcomes; Randomized Clinical Trial
MeSH Terms: conditions — Premature Birth; Brain Injuries; Leukomalacia, Periventricular | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO### (Placebo Comparator): All subjects will be identified as a such by the study identifier "EPO###" where EPO designates enrollment in this study and ### is a numeric identifier (e.g. 103).
  Interventions: Drug: Saline placebo
- EPO ### (Experimental): All subjects will be identified as a such by the study identifier "EPO###" where EPO designates enrollment in this study and ### is a numeric identifier (e.g. 103).
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — 5 of first 10 subjects (Group 1): 400 units/kg/dose once daily for 7 days 5 of next 10 subjects (Group 2): 800 units/kg/dose once daily for 7 days 20 of next 30 subjects (Group 3): 1000 units/kg/dose once daily for 7 days administered i.v. over 1 hour.
  The volume of the study drug will be 1 mL in a 1 mL Tuberculin syringe to be administered over 1 hour.
  Other Names: Confidential Randomization Number
  Arms: EPO ###
Drug: Saline placebo — Saline vehicle at a volume of 1 mL given over 1 hour intravenously once a day for the first seven days of life.
  Other Names: Confidential Randomization Number
  Arms: EPO###

SUMMARY:
The highest risk for perinatal brain injury occurs among extremely premature infants who weigh less than 1250 grams at birth. Such perinatal brain injury is currently irreversible, associated with neurodevelopmental disability, and without adequate treatment modalities. Research in recent years suggest in both animal and human studies that erythropoietin (Epo) may have significant neuroprotective effects. Given the historical safe medical profile of Epo when used for anemia of prematurity but the likely need for a greater dosage regimen for activation of neuroprotective pathways against neonatal brain injury, we therefore propose this phase II study of high-dose Epo in very low birth weight infants for the prevention and/or attenuation of prematurity-related cerebral hemorrhagic-ischemic injury.

DETAILED DESCRIPTION:
Eligible extremely premature infants will be enrolled in this double-blind, placebo-controlled randomized trial from the neonatal intensive care unit at Morristown Memorial Hospital (Morristown, New Jersey). Subjects will be enrolled within the first 24 hours of life and randomly assigned to receive Epo or saline vehicle placebo.

Standard NICU care will be provided to all subjects. Serial exams, CBC-d, reticulocyte counts, serum Epo levels, serial HUS, and head MRI will be collected at established time points during the study period. At 18 to 22 months corrected age, subjects will undergo a neurodevelopmental evaluation assessing for cerebral palsy, Bayley Scores of Infant Development-II (BSID-II) Mental Development Index (MDI), BSID-II Psychomotor Development Index (PDI), bilateral hearing aid use, and visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* 500 to 1250 grams at birth
* Less than 32 weeks gestation at birth
* Less than 24 hours of life at time of enrollment

Exclusion Criteria:

* Congenital anomalies (chromosomal, CNS, cardiac, GI, pulmonary)
* Seizures within first 24 hours of life
* Severe neutropenia (ANC < 500 cells/microL) within first 24 hours of life
* Polycythemia (Hct > 65%) within first 24 hours of life
* Thrombocytopenia (platelets < 50K cells/microL) within first 24 hours of life
* Hypertension (SBP > 100mmHg) without vasopressor support within first 24 hours of life

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental evaluations at 18 to 22 months corrected age (cerebral palsy, Bayley Scores of Infant Development Mental Development Index (MDI), Psychomotor Development Index (PDI), bilateral hearing aid use, and visual impairment) | 18-22 months corrected age

SECONDARY OUTCOMES:
Severe intraventricular hemorrhage | First ten days of life
Polycythemia, neutropenia, thrombocytopenia, hypertension, sepsis, hemorrhage, seizure | NICU hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

REFERENCES:
- [Background] Lin FK, Suggs S, Lin CH, Browne JK, Smalling R, Egrie JC, Chen KK, Fox GM, Martin F, Stabinsky Z, et al. Cloning and expression of the human erythropoietin gene. Proc Natl Acad Sci U S A. 1985 Nov;82(22):7580-4. doi: 10.1073/pnas.82.22.7580. PMID 3865178
- [Background] Ascensao JL, Bilgrami S, Zanjani ED. Erythropoietin. Biology and clinical applications. Am J Pediatr Hematol Oncol. 1991 Winter;13(4):376-87. doi: 10.1097/00043426-199124000-00002. PMID 1785666
- [Background] Buemi M, Aloisi C, Cavallaro E, Corica F, Floccari F, Grasso G, Lasco A, Pettinato G, Ruello A, Sturiale A, Frisina N. Recombinant human erythropoietin (rHuEPO): more than just the correction of uremic anemia. J Nephrol. 2002 Mar-Apr;15(2):97-103. PMID 12018644
- [Background] Fisher JW. Erythropoietin: physiology and pharmacology update. Exp Biol Med (Maywood). 2003 Jan;228(1):1-14. doi: 10.1177/153537020322800101. PMID 12524467
- [Background] Maier RF, Obladen M, Muller-Hansen I, Kattner E, Merz U, Arlettaz R, Groneck P, Hammer H, Kossel H, Verellen G, Stock GJ, Lacaze-Masmonteil T, Claris O, Wagner M, Matis J, Gilberg F; European Multicenter Erythropoietin Beta Study Group. Early treatment with erythropoietin beta ameliorates anemia and reduces transfusion requirements in infants with birth weights below 1000 g. J Pediatr. 2002 Jul;141(1):8-15. doi: 10.1067/mpd.2002.124309. PMID 12091844
- [Background] Ohls RK, Harcum J, Schibler KR, Christensen RD. The effect of erythropoietin on the transfusion requirements of preterm infants weighing 750 grams or less: a randomized, double-blind, placebo-controlled study. J Pediatr. 1997 Nov;131(5):661-5. doi: 10.1016/s0022-3476(97)70089-1. PMID 9403642
- [Background] Shannon KM, Keith JF 3rd, Mentzer WC, Ehrenkranz RA, Brown MS, Widness JA, Gleason CA, Bifano EM, Millard DD, Davis CB, et al. Recombinant human erythropoietin stimulates erythropoiesis and reduces erythrocyte transfusions in very low birth weight preterm infants. Pediatrics. 1995 Jan;95(1):1-8. PMID 7770284
- [Background] Meyer MP, Meyer JH, Commerford A, Hann FM, Sive AA, Moller G, Jacobs P, Malan AF. Recombinant human erythropoietin in the treatment of the anemia of prematurity: results of a double-blind, placebo-controlled study. Pediatrics. 1994 Jun;93(6 Pt 1):918-23. PMID 8190577
- [Background] Ohls RK, Ehrenkranz RA, Wright LL, Lemons JA, Korones SB, Stoll BJ, Stark AR, Shankaran S, Donovan EF, Close NC, Das A. Effects of early erythropoietin therapy on the transfusion requirements of preterm infants below 1250 grams birth weight: a multicenter, randomized, controlled trial. Pediatrics. 2001 Oct;108(4):934-42. doi: 10.1542/peds.108.4.934. PMID 11581447
- [Background] Brown MS, Keith JF 3rd. Comparison between two and five doses a week of recombinant human erythropoietin for anemia of prematurity: a randomized trial. Pediatrics. 1999 Aug;104(2 Pt 1):210-5. doi: 10.1542/peds.104.2.210. PMID 10428996
- [Background] Newton NR, Leonard CH, Piecuch RE, Phibbs RH. Neurodevelopmental outcome of prematurely born children treated with recombinant human erythropoietin in infancy. J Perinatol. 1999 Sep;19(6 Pt 1):403-6. doi: 10.1038/sj.jp.7200244. PMID 10685268
- [Background] Maier RF, Obladen M, Kattner E, Natzschka J, Messer J, Regazzoni BM, Speer CP, Fellman V, Grauel EL, Groneck P, Wagner M, Moriette G, Salle BL, Verellen G, Scigalla P. High-versus low-dose erythropoietin in extremely low birth weight infants. The European Multicenter rhEPO Study Group. J Pediatr. 1998 May;132(5):866-70. doi: 10.1016/s0022-3476(98)70320-8. PMID 9602202
- [Background] Shalak L, Perlman JM. Hemorrhagic-ischemic cerebral injury in the preterm infant: current concepts. Clin Perinatol. 2002 Dec;29(4):745-63. doi: 10.1016/s0095-5108(02)00048-9. PMID 12516744
- [Background] Guzzetta F, Shackelford GD, Volpe S, Perlman JM, Volpe JJ. Periventricular intraparenchymal echodensities in the premature newborn: critical determinant of neurologic outcome. Pediatrics. 1986 Dec;78(6):995-1006. PMID 3537951
- [Background] Bada HS, Green RS, Pourcyrous M, Leffler CW, Korones SB, Magill HL, Arheart K, Fitch CW, Anderson GD, Somes G, et al. Indomethacin reduces the risks of severe intraventricular hemorrhage. J Pediatr. 1989 Oct;115(4):631-7. doi: 10.1016/s0022-3476(89)80300-2. PMID 2677294
- [Background] Schmidt B, Davis P, Moddemann D, Ohlsson A, Roberts RS, Saigal S, Solimano A, Vincer M, Wright LL; Trial of Indomethacin Prophylaxis in Preterms Investigators. Long-term effects of indomethacin prophylaxis in extremely-low-birth-weight infants. N Engl J Med. 2001 Jun 28;344(26):1966-72. doi: 10.1056/NEJM200106283442602. PMID 11430325
- [Background] Juul S. Recombinant erythropoietin as a neuroprotective treatment: in vitro and in vivo models. Clin Perinatol. 2004 Mar;31(1):129-42. doi: 10.1016/j.clp.2004.03.004. PMID 15183662
- [Background] Wen TC, Rogido M, Genetta T, Sola A. Permanent focal cerebral ischemia activates erythropoietin receptor in the neonatal rat brain. Neurosci Lett. 2004 Jan 30;355(3):165-8. doi: 10.1016/j.neulet.2003.10.078. PMID 14732457
- [Background] Sola A, Rogido M, Lee BH, Genetta T, Wen TC. Erythropoietin after focal cerebral ischemia activates the Janus kinase-signal transducer and activator of transcription signaling pathway and improves brain injury in postnatal day 7 rats. Pediatr Res. 2005 Apr;57(4):481-7. doi: 10.1203/01.PDR.0000155760.88664.06. Epub 2005 Feb 17. PMID 15718373
- [Background] Sola A, Wen TC, Hamrick SE, Ferriero DM. Potential for protection and repair following injury to the developing brain: a role for erythropoietin? Pediatr Res. 2005 May;57(5 Pt 2):110R-117R. doi: 10.1203/01.PDR.0000159571.50758.39. Epub 2005 Apr 6. PMID 15817504
- [Background] Ehrenreich H, Hasselblatt M, Dembowski C, Cepek L, Lewczuk P, Stiefel M, Rustenbeck HH, Breiter N, Jacob S, Knerlich F, Bohn M, Poser W, Ruther E, Kochen M, Gefeller O, Gleiter C, Wessel TC, De Ryck M, Itri L, Prange H, Cerami A, Brines M, Siren AL. Erythropoietin therapy for acute stroke is both safe and beneficial. Mol Med. 2002 Aug;8(8):495-505. PMID 12435860
- [Background] Juul SE, Harcum J, Li Y, Christensen RD. Erythropoietin is present in the cerebrospinal fluid of neonates. J Pediatr. 1997 Mar;130(3):428-30. doi: 10.1016/s0022-3476(97)70205-1. PMID 9063419
- [Background] Brines ML, Ghezzi P, Keenan S, Agnello D, de Lanerolle NC, Cerami C, Itri LM, Cerami A. Erythropoietin crosses the blood-brain barrier to protect against experimental brain injury. Proc Natl Acad Sci U S A. 2000 Sep 12;97(19):10526-31. doi: 10.1073/pnas.97.19.10526. PMID 10984541
- [Background] Widness JA, Veng-Pedersen P, Peters C, Pereira LM, Schmidt RL, Lowe LS. Erythropoietin pharmacokinetics in premature infants: developmental, nonlinearity, and treatment effects. J Appl Physiol (1985). 1996 Jan;80(1):140-8. doi: 10.1152/jappl.1996.80.1.140. PMID 8847295
- [Background] Volpe JJ. Neurology of the newborn. 4th ed. Philadelphia: WB Saunders; 2001.